CLINICAL TRIAL: NCT05245266
Title: Improving Methods for Cell-Based Noninvasive Prenatal Testing (NIPT)
Brief Title: Cell-Based Noninvasive Prenatal Testing
Acronym: NIPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luna Genetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Luna IRB LG-003
Record Dates: First submitted 2022-02-03; First posted 2022-02-17 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy Related
Keywords: prenatal; genetic testing; noninvasive; diagnostic
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Analysis of blood samples from healthy pregnant women (Other): Analysis of blood samples from healthy pregnant women. A phlebotomist will be sent to any location in the United States to collect the blood sample. Sample identifiers will be removed as the first step so that laboratory personnel will not see or have access to identifiers. No information will go back to patients or their physicians.
  Interventions: Diagnostic Test: Redraw for analysis of blood samples from healthy pregnant women

INTERVENTIONS:
Diagnostic Test: Redraw for analysis of blood samples from healthy pregnant women — If less than two fetal cells are recovered from maternal blood, a redraw is indicated

SUMMARY:
The purpose of the overall study is to develop improved methods for recovery and analysis of fetal cells from the mother's blood in order to develop clinically useful forms of cell-based, diagnostic, noninvasive prenatal testing (NIPT). Luna genetics will obtain and analyze research blood samples from healthy pregnant women. A phlebotomist will be sent to any location in the United States to collect the blood samples. Sample identifiers will be removed as the first step so that laboratory personnel will not see or have access to identifiers.

ELIGIBILITY:
Inclusion Criteria for healthy pregnant subjects:

* Pregnant
* 18 years or older
* 65 or younger

Exclusion Criteria for healthy pregnant subjects:

* Acute illness
* Unavailability of maternal blood sample of at least 30 ml
* Language barrier (non-English speaking )
* Maternal age of less than 18 years, or over 65
* Higher order multiple pregnancy (triplet or greater)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All healthy pregnant female volunteers.
Enrollment: 500 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2024-01-12 (Estimated); Study Completion 2024-03-12 (Estimated)

PRIMARY OUTCOMES:
Number of fetal cells recovered and quality of DNA data on each cell | 3 years
  Outcome 1 is the number of cells identified as fetal by microscopic staining. This can be
  converted to units based on volume. If 40 mL of blood is collected and f8 cells are designated as fetal based on microscopic staining, the results can be tabulated as follow: So a result is 8 cells are identified as fetal from one blood draw. This equals 0.2 cells identified per mL of maternal blood. If two or fewer cells are obtained, a blood redraw will be requested from the patient.
Number of fetal cells recovered and quality of DNA data on each cell | 3 years
  Outcome measure 2 is the number of cells that yield high quality next generation
  sequencing data suitable for determining copy number across the entire genome. So if 4 of the 8 cells above gave high quality data, the outcome would be 4 cells with high quality copy number data from one blood draw which equals 0.10 high quality cell / mL of mother's b

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Beaudet, MD, Principal Investigator — Luna Genetics
Locations (1):
- Luna Genetics, Houston, Texas, United States